CLINICAL TRIAL: NCT00003144
Title: Phase I Study of Amifostine (Ethyol) as a Cytoprotector of Gemcitabine/Cisplatin Combination
Brief Title: Chemotherapy and Amifostine in Treating Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000065927; P30CA016087 (NIH); NYU-9722; ALZA-97-011-ii; NCI-V97-1363
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; drug/agent toxicity by tissue/organ
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Amifostine; Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the bad side effects of chemotherapy.

PURPOSE: Randomized phase I trial to study the effectiveness of amifostine in treating patients who are receiving chemotherapy for recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the ability of amifostine to facilitate increased dose escalation of gemcitabine and cisplatin. II. Compare the dose limiting toxicities of gemcitabine and cisplatin administered with and without amifostine in these patients. III. Determine the maximum tolerated dose of gemcitabine and cisplatin administered with amifostine in these patients. IV. Determine whether synergy is produced by administering gemcitabine and cisplatin on the same day.

OUTLINE: This is a two stage study. The first stage is a randomized study, and the second stage is a dose escalation study. In the first stage of the study, patients receive either intravenous gemcitabine/amifostine/cisplation (GAP) or gemcitabine/cisplatin (GP) in the first cycle. Patients are administered the other arm in the second cycle. In the second stage of the study (dose escalation), the initial dose of GP or GAP is given on days 1 and 8 every 28 days. Dose escalation is carried out in cohorts of 3 patients per dose level. If 1 of 3 patients experiences dose limiting toxicity (DLT), then 3 more patients are accrued at the same dose level. The maximum tolerated dose (MTD) is defined as the lowest dose at which 2 of 6 or 2 of 3 patients experience DLT. Patients experiencing grade 3 or 4 toxicity or tumor progression are removed from the study. Patients will be reassessed every 12 weeks.

PROJECTED ACCRUAL: A total of 32 patients will be accrued over 12-24 months in the first stage of this study, and 9-12 patients will be accrued for the second stage..

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory solid tumors Platinum sensitive

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: ECOG 0-2 Life Expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT less than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Other: No psychosis No significant medical illness No sensory neuropathy greater than grade 2

PRIOR CONCURRENT THERAPY: At least 3 weeks since prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 1997-08; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States